CLINICAL TRIAL: NCT06234826
Title: Skeletal Muscle Wasting in ICU Patients
Acronym: IC-MPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Frank Vandenabeele (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Sponsor-Investigator, Frank Vandenabeele, principal investigator, Hasselt University
Organization: Hasselt University (Other)
Other Study IDs: 2022/165
Record Dates: First submitted 2023-05-16; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Critical Illness; Muscle Atrophy
MeSH Terms: conditions — Critical Illness; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Muscle wasting occurs rapidly in critically ill patients and impacts both short and long term outcomes. Altered protein metabolism drives muscle loss in ICU patients, with muscle protein breakdown exceeding muscle protein synthesis (MPS). Interventions aimed at attenuating muscle loss by stimulating MPS rates are hampered by a lack of knowledge on altered muscle protein turnover rates during critical illness. Only a few studies have specifically assessed muscle protein synthesis by using contemporary intravenous stable isotope infusions, which allows the assessment of MPS over a short (<9 hours) period of time. Results from such acute studies can be difficult to extend or translate into long-term clinical practice and outcomes. Oral deuterated water (2H2O) dosing provides an alternative method that can be utilized to extend the measurement of muscle protein synthesis over a period of several days or weeks. It could therefore provide a valuable tool to study muscle protein synthesis during ICU admission and the impact of different anabolic interventions. Although multiple studies using the deuterated water methodology have been performed in both healthy volunteers and patients, it has not yet been performed in critically ill patients.

In this prospective study the investigators aim to assess fractional rates of muscle protein synthesis over a period of (maximal) 7 days in critically ill patients admitted to the intensive care unit. Secondly, the investigators aim to assess mechanisms of acute muscle wasting on an microscopic, ultrastructural and molecular level. Furthermore, the investigators aim to investigate to what extent muscle fibre size is recovered 3 months after ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* age >18y
* admitted to ICU
* enteral nutrition line in situ
* arterial line (any location) in situ
* expected stay ICU >7d

Exclusion Criteria:

* spinal cord injury
* chronic use of corticosteroids before hospital admission
* Contraindication to enteral infusion (e.g. due to GI-tract perforation)
* Kidney or liver failure
* therapeutic anti coagulation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In total 20 patients admitted to the ICU will be included.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
muscle protein synthesis rate (%/h) | 7 days of stay at the intensive care unit
  obtained by using deuterated water, muscle biopsy sampling and blood sampling

SECONDARY OUTCOMES:
skeletal muscle fiber characteristics 1 | 7 days of stay at the intensive care unit
  cross sectional area of muscle fibers
skeletal muscle fiber characteristics 2 | 7 days of stay at the intensive care unit
  amount and distribution of muscle fibers (distribution will be calculated as: amount of type X / total amount of fibres)
mRNA expression in skeletal muscle tissue 1 | 7 days of stay at the intensive care unit
  mRNA expression in skeletal muscle tissue of MAFBx (atrophy marker)
mRNA expression in skeletal muscle tissue 2 | 7 days of stay at the intensive care unit
  mRNA expression in skeletal muscle tissue of MurF1 (atrophy marker)
mRNA expression in skeletal muscle tissue 3 | 7 days of stay at the intensive care unit
  mRNA expression in skeletal muscle tissue of FOXO (atrophy marker)
patient characteristic- age | 7 days of stay at the intensive care unit
  age in years
patient characteristic- body weight | 7 days of stay at the intensive care unit
  body weight in kg
patient characteristic- height | 7 days of stay at the intensive care unit
  height in m
patient characteristic- sex | 7 days of stay at the intensive care unit
  male or female
patient characteristics (medical1) | 7 days of stay at the intensive care unit
  mechanical ventilation (duration in days)
patient characteristics (medical2) | 7 days of stay at the intensive care unit
  comorbidities (list of comorbidities)
patient characteristics (medical3) | 7 days of stay at the intensive care unit
  reason hospital admission
patient characteristic- APACHE score II | 7 days of stay at the intensive care unit
  APACHE II score = acute physiology score + age points + chronic health points. Minimum score = 0; maximum score = 71.
patient characteristic- food intake | 7 days of stay at the intensive care unit
  food intake (energy in kcal and protein intake in g/kg/d)
patient characteristic- LOS | Stay at the intensive care unit and Hospital (up to 1 year)
  Length of stay ICU and hospital (in days)
muscle volume | 3 months post-hospital discharge
  3d ultrasound assessed at follow up visit
habitual food | 3 months post-hospital discharge
  Assessed using questionnaires at follow up visit (higher score means better intake)
habitual activity | 3 months post-hospital discharge
  Assessed using questionnaires at follow up visit (higher score means better intake)
muscle hand grip strength | 3 months post-hospital discharge
  hand grip strength using the JAMAR dynamometer in kg
leg muscle strength | 3 months post-hospital discharge
  1RM upper leg at follow up visit
Functional capacity 1 | 3 months post-hospital discharge
  SPPB at follow up visit (short physical performance battery)
Functional capacity 2 | 3 months post-hospital discharge
  6min walking test at follow up visit
Quality of life questionnaire | 3 months post-hospital discharge
  SF-36 at follow up visit (Short Form Health Survey 36 items) range score between 0-100, lower score represents great health related problems
Quality of life questionnaires | 3 months post-hospital discharge
  Euro-QoL-5D-5-level at follow up visit (Euro quality of life 5 Dimension 5 level) Answers can be converted into EQ-5D index, an utility scores anchored at 0 for death and 1 for perfect health

CONTACTS AND LOCATIONS:
Overall Officials: Frank Vandenabeele, Prof., Principal Investigator — Hasselt University
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium